CLINICAL TRIAL: NCT06378931
Title: Quality of Life Change in Patients Undergoing Parathyroidectomy With Secondary Hyperparathyroidism Due to End-stage Renal Failure: a Prospective Cohort Study
Brief Title: Quality of Life Change in Patients Undergoing Parathyroidectomy With End-stage Renal Failure
Status: Not yet recruiting | Type: Observational
Sponsor: Chunling Jiang (Other)
Responsible Party: Sponsor-Investigator, Chunling Jiang, Professor, West China Hospital
Organization: West China Hospital (Other)
Other Study IDs: 2024HX161
Record Dates: First submitted 2024-03-26; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-03

CONDITIONS: Secondary Hyperparathyroidism; End Stage Renal Failure
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life change in patients Undergoing Parathyroidectomy with end-stage renal failure: Quality of Life Progression in Patients Undergoing Parathyroidectomy With Secondary Hyperparathyroidism Due to End-stage Renal Failure
  Interventions: Other: Quality of life progression after parathyroidectomy

INTERVENTIONS:
Other: Quality of life progression after parathyroidectomy — Study the progression of quality of life.

SUMMARY:
The purpose of this study is to characterize the quality of life change in patients undergoing parathyroidectomy with secondary hyperparathyroidism due to end-stage renal failure.

DETAILED DESCRIPTION:
Study participants will be asked questions about age, gender, education level, clinical symptoms, intensities of depression and anxiety, etc, and they will also be questioned regarding the prior quality of life score, as measured by the health-related quality of life 36-item Short-Form (SF-36) survey before surgery. Then, study participants will be contacted at one, three, six months, and 1 year after surgery, and asked questions about their SF-36 score, depression, and anxiety intensity.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old;
* Patients scheduled for parathyroidectomy with secondary hyperparathyroidism due to end-stage renal failure

Exclusion Criteria:

• Patients refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for parathyroidectomy with secondary hyperparathyroidism due to end-stage renal failure will be invited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-04-15 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Measure quality of life scores change with respect to time | up to 1 year
  Quality of life will be assessed by the 36-Item short form health survey scale, Subjects complete one response from a range of options for each of the 36 questions. A combination of item response is then aggregated to calculate a score for each of the eight dimensions listed. The scores for each dimension range from 0 to 100, with higher scores indicating better health status

SECONDARY OUTCOMES:
Measure anxiety and depression score change with respect to time | up to 1 year
  The anxiety and depression were evaluated using Hospital anxiety and depression Scale (HADS). The HADS consists of 14 questions, with 7 items each for the anxiety and depression subscales. The score for each item ranges from 0 to 3 points, and scores are summed to yield a separate score for anxiety (HADS-A) and depression (HADS-D).
Measure bone pain scores change with respect to time | up to 1 year
  The bone pain is evaluated using numerical rating scale (NRS). NRS scores range from 0 to 10 points, with 0 points representing no pain, 1-3 points representing mild pain, 4-6 points representing moderate pain, 7-9 points representing severe pain and 10 points representing the strongest pain.
Length of hospital stay | through study completion, an average of 1 week
  Determined by the number of days from admittance to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, Study Director — West China Hospital

IPD SHARING:
Plan to Share IPD: No